CLINICAL TRIAL: NCT06583083
Title: A Multicenter, Phase 2, Randomized Trial of Sintilimab (PD-1 Antibody) With P-GEMOX Versus the P-GEMOX Regimen in the Teatment of Newly Diagnosed Advanced-stage Extranodal Natural Killer/T Cell Lymphoma (ENKTL) (SPIRIT-02)
Brief Title: Sintilimab With P-GEMOX Versus the P-GEMOX in the Teatment of Advanced-stage Extranodal Natural Killer/T Cell Lymphoma
Acronym: SPIRIT-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-475-01
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
MeSH Terms: interventions — sintilimab; pegaspargase; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Sintilimab with P-GEMOX Regimen
  Interventions: Drug: Sintilimab with P-GEMOX Regimen
- control group (Active Comparator): P-GEMOX Regimen
  Interventions: Drug: P-GEMOX Regimen

INTERVENTIONS:
Drug: Sintilimab with P-GEMOX Regimen — Sintilimab intravenous drip, Pegaspargase intramuscular injection, gemcitabine intravenous drip, oxaliplatin intravenous drip
  Other Names: Sintilimab, Pegaspargase, gemcitabine, oxaliplatin
  Arms: experimental group
Drug: P-GEMOX Regimen — Pegaspargase intramuscular injection, gemcitabine intravenous drip, oxaliplatin intravenous drip
  Other Names: Pegaspargase, gemcitabine, oxaliplatin
  Arms: control group

SUMMARY:
Extranodal NK/T-cell lymphoma is a rare and highly aggressive subtype of non-Hodgkin lymphoma. While the overall survival rates have improved for early-stage ENKTL patients, the prognosis for those with advanced disease remains poor, and there is currently no standard treatment. PD-1/PD-L1 inhibitors have demonstrated significant efficacy in various cancers, and recent studies have shown promising results in extranodal NK/T-cell lymphoma as well. Although PD-1 antibodies have exhibited efficacy in relapsed or refractory patients, their effectiveness when combined with chemotherapy as a first-line treatment remains unclear. This study aims to evaluate the efficacy and safety of sintilimab combined with chemotherapy in a randomized controlled trial for newly diagnosed advanced extranodal NK/T-cell lymphoma patients, while also exploring potential biomarkers that may predict treatment outcomes, offering new therapeutic options for extranodal NK/T-cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with ENKTL.
2. Advanced stage.
3. Has at least one measurable or assessable lesion.
4. Age > 18 years, no gender restrictions, with an expected survival of more than 3 months.
5. Willing to participate in the clinical study; fully informed and has signed a written informed consent form.
6. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Aggressive NK-cell leukemia.
2. Central nervous system involvement.
3. Patients with significant dysfunction of vital organs.
4. History of allergy to the investigational drug, similar drugs, or excipients.
5. Less than 6 weeks since major organ surgery (excluding surgery for biopsy purposes).
6. Pregnant or breastfeeding women, and women of childbearing potential who are unwilling to use contraception.
7. Active infection, excluding fever related to tumor-associated B symptoms.
8. Known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome (AIDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 4 years
  progression free survival

SECONDARY OUTCOMES:
ORR rate | Up to 4 years
  objective response rate
CR rate | Up to 4 years
  complete response rate
OS | Up to 4 years
  overall survival
Adverse events | Up to 4 years
  The incedence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Guangzhou, Guangdong, China